CLINICAL TRIAL: NCT05304832
Title: The Effectiveness of Aqua-plyometric Exercises for Muscle Strength, Bone Health, and Physical Ability in Patients With Juvenile Idiopathic Arthritis. A 12-week, Randomized Controlled Trial
Brief Title: The Role of Aquatic-Based Plyometric Exercises for Patients With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ragab Kamal Elnaggar, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RHPT/0020/0045
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Intervention Model Description: A prospective, dual-arm, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: This was a single-blind protocol. The researcher who collected the data was blind to the allocation of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AquaPlyo group (Experimental): Participants in this group received the AquaPlyo training program
  Interventions: Other: Aqua-Plyometric Exercise
- Control group (Active Comparator): Participants in this group received the standard exercise program.
  Interventions: Other: Standard physical therapy

INTERVENTIONS:
Other: Aqua-Plyometric Exercise — The aqua-plyometric training was conducted for 45 minutes, twice weekly, for 12 successive weeks. The training was geared toward the lower body and was conducted under close supervision of a licensed pediatric physical therapist in accordance with the safety performance guidelines defined by the American Academy of Pediatrics and the US National Strength and Conditioning Association.
  Arms: AquaPlyo group
Other: Standard physical therapy — The program encompassed the standard exercises for patients with JIA (aerobic, weight-bearing, proprioceptive, flexibility, and strengthening exercises). The training was conducted for 40 minutes, two times a week for 12 successive weeks.
  Arms: Control group

SUMMARY:
This study was designed to assess the effect of a 12-week aqua-plyometric (AquaPlyo) training on muscle strength, bone health, and physical ability in children with juvenile idiopathic arthritis (JIA). Forty-eight patients with JIA were randomly allocated to the AquaPlyo group (n = 24, received an aquatic-based plyometric training program, twice/week, over 12 weeks) or the control group (n = 24, received standard exercise program). Both groups were assessed for muscle strength, bone health, and physical ability pre and post-treatment.

DETAILED DESCRIPTION:
Forty-eight patients with JIA were recruited from the pediatric rheumatology clinics of three large referral hospitals in Riyadh, Saudi Arabia. The study included patients who had a confirmed diagnosis of Polyarticular JIA (according to the criteria set forth by the International League of Associations for Rheumatology), aged 12-18 years, identified being stable cases, and did not participate in a regular exercise program (in the past six months). Patients who had fixed deformities, a history of joint surgery, or whose radiological investigations revealed erosive changes of bone, ankylosing, or fractures were excluded.

Outcome measures

1. Muscle strength: The peak concentric torque of the right and left quadriceps muscle was measured through an Isokinetic Dynamometer.
2. Bone health: Areal bone mineral density, volumetric bone density, and bone mineral content of the lumbar spine and neck of femur were measured through Dual-Energy X-ray Absorptiometry (DEXA) scanning.
3. Physical ability: The physical performance was assessed using the 6-minute walk test.

The AquaPlyo group received a 12-week AquaPlyo training, 45 minutes per session, two times a week for 12 consecutive weeks, in conformity with the National Strength and Conditioning Association guidelines and American Academy of Pediatrics safety standards. The AquaPlyo program consisted of ten unilateral and bilateral lower limb plyometrics in the form of hopping/bounding/jumping activities conducted in a water medium. The AquaPlyo training included a warm-up for 10 minutes and a cool-down for 5 minutes. The control group received the standard exercise program, 45 minutes per session, two times a week for 12 consecutive weeks. The program consisted of flexibility exercise, strength training, weight-bearing, proprioceptive training, and free treadmill walking or cycle ergometry.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of JIA
* Polyarticular onset of JIA with bilateral involvement of the knee joint
* Age between 12 and 18 years
* Stable conditions (i.e., receive stable doses of medications in the past three months)
* Not participating in a regular exercise program in the past six months

Exclusion Criteria:

* Fixed deformities
* History of joint surgery
* Ankylosing or fractures
* Bone destruction (erosive changes of the knee joint)
* Cardiopulmonary comorbidities
* Recommendation against engaging in potentially explosive physical activities by the attending Rheumatologist.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-06 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 2 months
  Indicated by the peak concentric torque of the quadriceps muscle (Nm). It was measured using an Isokinetic Dynamometer.
Areal bone mineral density | 2 months
  The amount of bone mineral divided by the bone scanned area (gm/cm2). It was assessed through DEXA scanining.
Volumetric bone mineral density | 2 months
  The mineral mass per unit volume of bone (gm/cm3). It was assessed through DEXA scanining.
Bone mineral content | 2 months
  It is the amount of bone mineral in bone tissue (g/cm). It was calculated by summing the bone mineral density values over the projected area.

SECONDARY OUTCOMES:
Physical ability | 2 months
  The maximum distance (m) that participants were able to cover during the 6-minute walk test.

CONTACTS AND LOCATIONS:
Overall Officials: Ragab K Elnaggar, PhD, Principal Investigator — Prince Sattam Bin Abdulaziz University
Locations (1):
- Ragab K. Elnaggar, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elnaggar RK, Elfakharany MS. Aqua-Plyometric Exercises-Induced Changes in Muscle Strength, Bone Mineral Properties, and Physical Fitness in Patients With Juvenile Idiopathic Arthritis: A 12-Week, Randomized Controlled Trial. Pediatr Exerc Sci. 2022 Dec 19;35(4):198-205. doi: 10.1123/pes.2022-0044. Print 2023 Nov 1. PMID 36535274